CLINICAL TRIAL: NCT02572531
Title: Effect of Probiotic Supplements on Pain and Oral Wound Healing After Third Molar Surgery
Brief Title: Effect of Probiotics on Pain and Oral Wound Healing After Third Molar Surgery
Acronym: PROVIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Copenhagen (Other)
Collaborators: Halmstad County Hospital (Other)
Responsible Party: Principal Investigator, Gina Castiblanco, Dr., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2015-483
Record Dates: First submitted 2015-09-14; First posted 2015-10-09 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Complications
Keywords: Lactobacillus reuteri; Wound Healing; Third Molar; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri (Active Comparator): L. reuteri DSM 17938/ATCC PTA L. reuteri DSM 17938/ATCC PTA lozenges three times daily for 2 weeks
  Interventions: Dietary Supplement: L. reuteri DSM 17938/ATCC PTA
- Placebo (Placebo Comparator): Placebo lozenges three times daily for 2 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938/ATCC PTA — Ingestion of active lozenge three times daily for 2 weeks
  Arms: L. reuteri
Dietary Supplement: Placebo — Ingestion of placebo lozenge three times daily for 2 weeks
  Arms: Placebo

SUMMARY:
The aim of this research is to study the effect of probiotic supplements (Lactobacillus reuteri) on post-surgical complications and oral wound healing after extraction of impacted third molars.

DETAILED DESCRIPTION:
Healthy volunteers are consecutively randomized to the test or placebo group. After a standardized surgical procedure, conducted under local anesthesia, the participants are instructed to take three lozenges daily (one in the morning, one at lunch time and one in the evening) containing either two strains of L. reuteri (DSM 17938 and ATCC PTA 5289; >108 CFU per lozenge) or placebo for 2 weeks. The subjects are instructed to let the tablet slowly melt in the oral cavity and to fill in a personal log-book on a daily basis throughout the postoperative period. The patients are recalled to the clinic for follow-up after 1, 2 and 3 weeks for examination. The post-surgical events (pain, swelling, discomfort, feeding problems) are registered daily by the patient in a custom-made logbook. Furthermore, the type and frequency of painkillers and antibiotic prescriptions are noted in the logbook. At the follow-ups, the healing of the wounds/lesions is scored with a clinical healing index. Stimulated saliva samples are collected at baseline and after 2 weeks and kept frozen until further analysis. In addition, smear samples are collected after 1 and 2 weeks from the extraction socket for bacterial analysis. Any subjectively perceived side- or adverse effect in connection with the intervention should be reported to the surgeon. The participants are encouraged to maintain their normal tooth brushing habits.

ELIGIBILITY:
Inclusion Criteria:

* Uncompromised general health
* Non-smoker
* No systemic medications (except contraceptives)
* No recent/ongoing episode of antibiotic treatment.

Exclusion Criteria:

* Any pathological condition associated with the third molars detected on radiographs prior to surgery
* Regular consumers of probiotics

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain with VAS scale (0-10) | Three weeks: Baseline and 3 follow ups
  VAS scale of the patient's perception of pain (0- I don´t feel any pain, 10- unbearable pain)
Change from Baseline in Swelling with VAS scale (0-10) | Three weeks: Baseline and 3 follow ups
  VAS scale of the patient's perception of swelling (0- not swollen at all, 10- extremely swolen, can hardly swallow)
Change from Baseline in Feeding Problems with VAS scale (0-10) | Three weeks: Baseline and 3 follow ups
  VAS scale of the patient's perception of feeding problems related to the surgery (0- I eat as usual, 10- hardly eat/liquid food ingestion)
Change from Baseline in Discomfort with VAS scale (0-10) | Three weeks: Baseline and 3 follow ups
  VAS scale of the patient's perception of discomfort (0- No discomfort at all, 10- high discomfort-can not perform daily activities)
Frequency of Painkillers Intake after Surgery | Three weeks: Baseline and 3 follow ups
  Frequency expressed in number of painkillers taken per day
Frequency of Antibiotics Intake after Surgery | Three weeks: Baseline and 3 follow ups
  Frequency expressed in number of antibiotics taken per day

SECONDARY OUTCOMES:
Clinical healing index by Landry et al. Scale from 1-5 (1 very poor healing - 5 very good healing) | Three weeks: 3 follow-ups
  Healing index by Landry et al. Scale from 1-5 (1 very poor healing - 5 very good healing) assessed by the maxillofacial surgeon
Levels of salivary oxcytocin | Two weeks: Baseline and two weeks after surgery
Microbial counts | Two weeks: First and Second Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Svante Twetman, Professor, Study Director — University of Copenhagen

REFERENCES:
- [Background] Poutahidis T, Kearney SM, Levkovich T, Qi P, Varian BJ, Lakritz JR, Ibrahim YM, Chatzigiagkos A, Alm EJ, Erdman SE. Microbial symbionts accelerate wound healing via the neuropeptide hormone oxytocin. PLoS One. 2013 Oct 30;8(10):e78898. doi: 10.1371/journal.pone.0078898. eCollection 2013. PMID 24205344